CLINICAL TRIAL: NCT06052397
Title: Sleep and Circadian Rhythm Biomarkers of Postoperative Delirium
Acronym: SLEEP-POD
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lei Gao, MBBS, MMSc, Attending Physician, Department of Anesthesia, Critical Care, and Pain Medicine, Massachusetts General Hospital
Other Study IDs: 2023P000596
Record Dates: First submitted 2023-08-21; First posted 2023-09-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Delirium, Postoperative; Cognitive Decline; Dementia
Keywords: Sleep; Postoperative Delirium; Circadian Rhythms; Cognition; Dementia
MeSH Terms: conditions — Emergence Delirium; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sleep and Circadian Rhythms biomarker cohort: Cohort will complete a series of blood sample donations (both intraoperatively and postoperatively) as well as complete daily neurocognitive assessments at baseline and on PODs 1 - 3.

SUMMARY:
The goal of this prospective cohort study is to assess potential differences in sleep biomarkers in older adult patients undergoing major orthopedic surgery. The main questions it aims to answer are:

1. To define sleep/circadian biomarkers of delirium (sleep duration, regularity, stability and timing of rhythm) in a prospective observational study.
2. To determine if plasma Alzheimer's disease (AD) pathology/inflammatory burden interacts with or moderates the relationship between a sleep/circadian biomarker and post-operative delirium (POD) risk.
3. To determine whether sleep/circadian regulation interacts with the genetic risk of AD to influence POD/cognitive decline.

Participants will be asked to:

1. Donate several blood samples both intraoperatively and postoperatively
2. Complete baseline and postoperative neurocognitive assessments
3. Wear an actigraphy data collection watch for the two weeks prior to their surgery

DETAILED DESCRIPTION:
This study is a prospective, observational study designed to identify changes in protein biomarkers levels as a function of delirium incidence and delirium severity scores based on Confusion Assessment Method (CAM) scores from postoperative days 1-3. Additionally, patients will wear an Actiwatch to monitor sleep/circadian rhythm biomarkers. Questionnaires gathering information about sleep, cognition, mood, pain, and physical/social function will be asked throughout the course of the study. There is no intervention being tested in this study. Accepted standard of care involving all clinical procedures, pain management, and anesthesia and surgical care, will be performed within this study. Patients will be contacted remotely at 1-month, 3-months, and 12-months for follow-up visits that will include questionnaires and actigraphy assessments.

If possible, the patient will be enrolled in person where the member of the study team will complete all enrollment procedures if time allows. The baseline procedures will include fitting the Actiwatch, going over Actiwatch usage instructions, and a baseline neurocognitive assessment and questionnaires. If there is not enough time for complete these procedures, or if the patient is approached over the phone, a member of the study team can complete these baseline procedures with the patient remotely. Baseline assessments can be completed over the phone, and the Actiwatch will be mailed directly to the patient's preferred address.

Clinical Data Collection - Clinical data but not limited to including age, sex, body mass index (BMI), length of hospital stay, and surgical details (e.g., surgery duration, anesthesia type, blood loss, complications) will be recorded using passively collected data from the patient's electronic medical record. Information about history of sleep, cognition/neurology, psychiatry, pain management, and physical/social function that cannot be inferred from the patient's medical record will be elicited from the participant directly at the time of the baseline questionnaires.

Actiwatch Data Collection - Patients will wear the Actiwatch continuously for at least seven days but no more than two weeks leading up to surgery. The watch will be distributed with a specific instruction sheet, and the study team will ensure that all questions have been answered. Patients who are consented at the time of their preoperative clinic visit will be given their watch at the time of their appointment. For patients who are consented virtually, the watch will be mailed to their preferred home address. The watch will collect data including sleep duration, regularity, stability and timing of rhythm. Patients will return the watch on the day of surgery. Patients will be asked to wear the watch for one week at the time of their 1-, 3-, and 12-month timepoints as well. Watches will be returned to the participant via mail and a prepaid mailing envelope will be sent with the watch so that the patient can return it at the conclusion of the recording period.

Sleep Diary - Patients will be asked to fill out a sleep diary on the days that they wear the Actiwatch. The diary will ask questions regarding their sleep habits and factors that might affect their ability to fall asleep. The sleep diary should be filled out during the period leading up to the patient's surgery and again at their 1-, 3-, and 12-month follow-up visits.

ECG Data Collection - Electrocardiogram data will be collected using a 4-lead ECG monitor with oximetry. During the inclusion visit, a study staff member will fit the ECG and oximeter to the patient and record for 30 minutes. The device can connect to an app for Bluetooth ECG reading display. Study staff will monitor the live recording to ensure that data is being collected accurately. The ECG-oximetry data can provide information about cardio physiological biomarkers for delirium. This study measure can be taken either at the time of consent (for patients who consent in-person), or in the preoperative holding area on the day of surgery. An additional recording will occur for 30 minutes perioperatively. If either ECG recording cannot be performed, this will not be considered a protocol deviation.

EEG Data Collection - If the anesthesiologist places a SedLine for EEG for clinically-indicated surface level electroencephalogram monitoring while the patient is under general anesthesia, a study staff member may record the data to be used later to explore EEG biomarkers of delirium risk. If the EEG recording cannot be collected, this will not be considered a protocol deviation.

Assessments - The Montreal Cognitive Assessment (MoCA) will be performed during the baseline visit at the preoperative clinic site, or over the phone using the telephonic version (tMoCA). The MoCA will also be completed daily on postoperative days 1, 2, and 3. The long-form of the Confusion Assessment Method (CAM) will be performed at the baseline visit or baseline phone-call and twice daily on postoperative days 1 through 3 (morning and afternoon). In the afternoons during the first three days postoperatively, a standard cognitive assessment will be performed in order to appropriately score the CAM. The postoperative assessments will be performed by a trained member of the study team. The tMoCA will be completed at the 1-month, 3-month, and 12-month follow up periods.

The CAM-long form will be applied twice daily from preoperative day 1 to postoperative day 3 to evaluate cognitive changes in each patient, and the peak delirium severity score will be used for comparative analyses. CAM scores will be recorded for each patient to determine if the criteria for a positive delirium screen have been met. The Montreal Cognitive Assessment (MoCA) will also be used to evaluate cognitive differences at baseline during the preoperative evaluation.

Additionally, subjects will complete sleep disturbance questionnaires at the time of their baseline visit and at 1-, 3-, and 12 months after surgery including the Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI), Epworth Sleepiness Scale (ESS), and a chronotype questionnaire (only asked at baseline). The Geriatric Depression Scale (GDS) and Generalized Anxiety Disorder 7 (GAD-7) questionnaires will be administered to gather information about the patient's mood. The PROMIS Pain Interference Short Form questionnaire and a Verbal Rating Scale will be used to assess pain experienced by the patients. The Functional Activities Questionnaire (FAQ), FRAIL Scale, and UCLA Loneliness Scale will be administered to assess physical and social function of the patient. These questionnaires can be administered at any point during the baseline and 1-month, 3-month, and 12-month follow-up periods (4 administrations, 1 at each period) at the hospital, over the phone, or via a secure REDCap survey patients can fill out remotely.

Patients will be contacted over the phone or through email across the course of participation to clarify study procedures and to coordinate virtual follow-up visits as necessary.

To assess for the impact of nutrition on the collected blood samples, a nutrition assessment will be performed prior to blood collection.

Details regarding patient-centered clinical outcomes, including delirium onset, delirium severity, mortality, and hospital length of stay, will be collected using our electronic medical record.

Blood Collection:

First blood draw (20ml): Preoperative day 0 (0-2 hours before surgery)

Second blood draw (10ml): Postoperative day 1 (± 1 day)

When possible, blood collection will be performed while the patient is under general anesthesia and be extracted from an indwelling line to minimize patient discomfort. Trained study staff may perform the phlebotomy, but we will not consider it a protocol deviation if blood cannot be collected due to insufficient staff training, IV availability, or patient refusal. A one-day window will be employed for the postoperative assessment to enhance collection efforts if a sample cannot be obtained on postoperative day one.

Targeted protein screens and metabolomics analysis will then be used to analyze blood to determine the relative metabolic and inflammatory protein abundance and steady-state metabolite levels at each timepoint.

Coded Samples: All blood samples will be assigned a unique sample ID, containing no identifiers that can be associated with the subject. The sample ID will be used for all data analysis and provided to the core facilities for analyses. The sample ID and associated patient MRN crosswalk will be stored in a secure and locked spreadsheet and only available to the MGB IRB-approved study team.

Sample Processing: Whole-blood samples will be collected and immediately processed for plasma and DNA isolation in the laboratory. Briefly, blood collected preoperatively will be transferred to a plasma and buffy coat separator tube with clot factor (EDTA - purple top tube), followed by centrifugation at 3000rpm for 30 minutes. The supernatant (plasma) and buffy coat (DNA) will then be collected, aliquoted, and stored at -80°C until further processing. Blood collected postoperatively will be transferred to a plasma separator tube with clot factor (NA citrate - blue top tube), followed by centrifugation at 3000rpm for 30 minutes. The supernatant (plasma) will then be collected, aliquoted, and stored at -80°C until further processing.

Genetic Analysis from Blood Samples: To gather information about AD variant genes, including APOE-ε4, we may send the coded blood samples for genotyping in-house at the MGH Center for Computational and Integrative Biology (per their published Mass General Brigham Members Genotyping rates). Results regarding the genotypic data will be securely stored in encrypted and password-protected devices per MGB requirements. No personal identifiers will be shared. Participants will not be made aware of their AD gene risk status.

Rigor and Reproducibility: The clinical study will follow institutional and federal guidelines for clinical research. All delirium assessments will be conducted by trained researchers. All source documents will be securely stored in encrypted and password protected devices in accordance with MGB requirements.

These study procedures will allow us to complete data analysis towards our objective of investigating the impact of sleep/circadian disruption on POD risk by defining the preoperative and postoperative profile of amyloid, tau, and neurodegeneration (ATN) biomarkers and proteomic signatures (inflammatory and metabolic) in older patients undergoing major non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 70 years old
* Scheduled to undergo major orthopedic surgery
* Expected postoperative recovery of more than 24 hours as an inpatient

Exclusion Criteria:

* Cognitive impairment leading to inability to consent
* Patients with limited mobility or inability to wear an actigraphy watch
* Patients with infection at the site of actigraphy watch, allergies to materials of watch
* Patients with > two days in the ICU during the month prior to surgery
* Renal or liver failure
* Severe neurocognitive damage or history of psychiatric illness
* Blindness or deafness
* Patients who are non-English speaking

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The Targeted/Planned enrollment for the proposed clinical study is consistent with the ethnic and racial composition of Suffolk County, MA. Please see below.
  American Indian and Alaska Native - 0.7 Native Hawaiian and Other Pacific Islander - 0.2 Asian - 9.3 Black, not Hispanic or Latino - 24.3 White, not Hispanic or Latino - 45.2 Hispanic or Latino - 23.3 Two or more races - 3.7 Female - 51.7
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Delirium | From postoperative day 1 to postoperative day 3
  Outcome will be assessed using the Confusion Assessment Method (CAM)

SECONDARY OUTCOMES:
Severity of Delirium | From postoperative day 1 to postoperative day 3
  CAM: Minimum Score=0, Maximum Score=19, Higher Scores: indicate increased severity of delirium
Delirium-free Days | Up until postoperative day 3, or up until postoperative day 7 or discharge for patients who are delirious beyond postoperative day 5
  CAM
Postoperative Cognitive Status | Months 1, 3, and 12 after surgery
  Telephone Montreal Cognitive Assessment (tMoCA): Minimum Score=0, Maximum Score=22, Higher Scores: indicate better cognitive function
Postoperative Insomnia Symptom Severity | Baseline and months 1, 3, and 12 after surgery
  Insomnia Severity Index, with lower scores being considered better
Postoperative Sleep Quality | Baseline and months 1, 3, and 12 after surgery
  Pittsburgh Sleep Quality Index, with lower scores being considered better
Postoperative Sleepiness | Baseline and months 1, 3, and 12 after surgery
  Epworth Sleepiness Scale, with lower scores being considered better.
Postoperative Depression | Baseline and months 1, 3, and 12 after surgery
  Assessed via Geriatric Depression Scale with lower scores being considered better.
Postoperative Anxiety | Baseline and months 1, 3, and 12 after surgery
  Assessed via Generalized Anxiety Disorder - 7 with lower scores being considered better
Postoperative Physical Function | Baseline and months 1, 3, and 12 after surgery
  Functional Activities Questionnaire with lower scores being better
Postoperative Physical Frailty | Baseline and months 1, 3, and 12 after surgery
  FRAIL Scale with lower scores being better
Postoperative Social Function | Baseline and months 1, 3, and 12 after surgery
  UCLA Loneliness Scale with lower scores being better
Blood Delirium Biomarkers - IL-6 | Day of surgery up until postoperative day 3
  Blood samples including whole blood and serum will be collected to define the pre and post-operative profiles of IL-6 biomarkers
Blood Delirium Biomarkers - C-reactive protein | Day of surgery up until postoperative day 3
  Blood samples including whole blood and serum will be collected to define the pre and post-operative profiles of C-reactive protein biomarkers
Blood Delirium Biomarkers - Tau-PT181 | Day of surgery up until postoperative day 3
  Blood samples including whole blood and serum will be collected to define the pre and post-operative profiles of Tau-PT181 biomarkers
Blood Delirium Biomarkers - Tau-PT217 | Day of surgery up until postoperative day 3
  Blood samples including whole blood and serum will be collected to define the pre and post-operative profiles of Tau-PT217 biomarkers

OTHER OUTCOMES:
Length of Hospital Stay | Date of hospital admission up until date of discharge, assessed up to 30 days
  Medical Record Review

CONTACTS AND LOCATIONS:
Overall Officials: Lei Gao, MBBS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient specimens and data may be shared with individuals who are members of the IRB-approved research team or approved for sharing within the MGB network.
Supporting Information: Study Protocol, SAP
Time Frame: Data may be shared with collaborators once the study has been completed.
Access Criteria: IRB approved research team members or approved collaborators within MGB.

REFERENCES:
- [Background] Ulsa MC, Xi Z, Li P, Gaba A, Wong PM, Saxena R, Scheer FAJL, Rutter M, Akeju O, Hu K, Gao L. Association of Poor Sleep Burden in Middle Age and Older Adults With Risk for Delirium During Hospitalization. J Gerontol A Biol Sci Med Sci. 2022 Mar 3;77(3):507-516. doi: 10.1093/gerona/glab272. PMID 34558609
- [Background] Dessap AM, Roche-Campo F, Launay JM, Charles-Nelson A, Katsahian S, Brun-Buisson C, Brochard L. Delirium and Circadian Rhythm of Melatonin During Weaning From Mechanical Ventilation: An Ancillary Study of a Weaning Trial. Chest. 2015 Nov;148(5):1231-1241. doi: 10.1378/chest.15-0525. PMID 26158245
- [Background] Miner B, Kryger MH. Sleep in the Aging Population. Sleep Med Clin. 2017 Mar;12(1):31-38. doi: 10.1016/j.jsmc.2016.10.008. Epub 2016 Dec 20. PMID 28159095
- [Background] American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults. Postoperative delirium in older adults: best practice statement from the American Geriatrics Society. J Am Coll Surg. 2015 Feb;220(2):136-48.e1. doi: 10.1016/j.jamcollsurg.2014.10.019. Epub 2014 Nov 14. No abstract available. PMID 25535170
- [Background] Gou RY, Hshieh TT, Marcantonio ER, Cooper Z, Jones RN, Travison TG, Fong TG, Abdeen A, Lange J, Earp B, Schmitt EM, Leslie DL, Inouye SK; SAGES Study Group. One-Year Medicare Costs Associated With Delirium in Older Patients Undergoing Major Elective Surgery. JAMA Surg. 2021 May 1;156(5):430-442. doi: 10.1001/jamasurg.2020.7260. PMID 33625501
- [Background] Rahman S, Byatt K. Follow-up services for delirium after COVID-19-where now? Age Ageing. 2021 May 5;50(3):601-604. doi: 10.1093/ageing/afab014. PMID 33951153
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] O'Gara BP, Gao L, Marcantonio ER, Subramaniam B. Sleep, Pain, and Cognition: Modifiable Targets for Optimal Perioperative Brain Health. Anesthesiology. 2021 Dec 1;135(6):1132-1152. doi: 10.1097/ALN.0000000000004046. PMID 34731233
- [Background] Gao L, Li P, Gaykova N, Zheng X, Gao C, Lane JM, Saxena R, Scheer FAJL, Rutter MK, Akeju O, Hu K. Circadian Rest-Activity Rhythms, Delirium Risk, and Progression to Dementia. Ann Neurol. 2023 Jun;93(6):1145-1157. doi: 10.1002/ana.26617. Epub 2023 Mar 3. PMID 36808743
- [Derived] Sugg E, Gleeson E, Baker SN, Li P, Gao C, Mueller A, Deng H, Shen S, Franco-Garcia E, Saxena R, Musiek ES, Akeju O, Xie Z, Hu K, Gao L. Sleep and circadian biomarkers of postoperative delirium (SLEEP-POD): protocol for a prospective and observational cohort study. BMJ Open. 2024 Apr 19;14(4):e080796. doi: 10.1136/bmjopen-2023-080796. PMID 38643014